CLINICAL TRIAL: NCT00528294
Title: Phase I Trial From GRID 18F-FDG-PET Biological Imaging-guided Intensitymodulated Radiotherapy (BG-IMRT) With Patients With Recurrent or New Head or Neck Tumor in Previously Radiated Area
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study status unknown Investigator retired and no longer working in the institution.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/010
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2014-12

CONDITIONS: Head and Neck Tumors
Keywords: Recurrent head and neck tumors
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): GRID-radiotherapy followed by biological imaging guided IMRT
  Interventions: Radiation: GRID radiotherapy

INTERVENTIONS:
Radiation: GRID radiotherapy — GRID-radiotherapy followed by biological imaging guided IMRT

SUMMARY:
This trials examines the feasibility of GRID-therapy combined with biologically imaging based IMRT (BG-IMRT). Within this trial, the strict toxicity parameters of primary treatment of head and neck tumors are used. The GRID and BG-IMRT technique might be possible to reduce the total radiation dose 2 to 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or new head or neck tumor
* 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose. | 3 months after end of treatment
Superior local control with Grid 18F-FDG-PET BG-IMRT using previously obtained maximum tolerated dose. | 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be